CLINICAL TRIAL: NCT00690300
Title: Phase II Study: Docetaxel Plus Oxaliplatin as Second-line Therapy in Patients With Advanced Metastatic Pancreatic Cancer
Brief Title: Docetaxel Plus Oxaliplatin as Therapy in Patients With Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Prof. Dr. Thomas Seufferlein, University Halle-Wittenberg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I1-GOA-1; EudraCT 2005-004236-40
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-01

CONDITIONS: Pancreas Neoplasms
Keywords: adenocarcinoma of the pancreas; pancreatic cancer; pancreas carcinoma; advanced pancreatic cancer; metastatic pancreatic cancer; second line; palliative; Oxaliplatin; Docetaxel; Taxotere; Eloxatin; Cancer of pancreas; Pancreas cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Docetaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 IV on day 1 of each 22 day cycle
  Other Names: Taxotere
Drug: Oxaliplatin — 80 mg/m2 IV on day 2 of each 22 day cycle
  Other Names: Eloxatin

SUMMARY:
The purpose of this study is to test a combination-therapy of oxaliplatin and docetaxel in patients with metastatic or locally advanced adenocarcinoma of the pancreas after failure of a palliative first line therapy.

DETAILED DESCRIPTION:
For years Fluorouracil was the established treatment for pancreatic cancer with median survival times up to 8 months. Since 1997 Gemcitabine is also a standard therapy with in comparison to Fluorouracil a significant better clinical benefit.

But after progression of the disease under a palliative first-line therapy there is no established second line therapy for pancreatic cancer.

So the purpose of this study is to test the combination of Oxaliplatin and Docetaxel in patients with metastatic or locally advanced adenocarcinoma of the pancreas after failure of a palliative first line therapy to get a reasonable second line concept.

ELIGIBILITY:
Inclusion Criteria:

* Dated and signed informed concent
* Histologically or cytologically proven metastatic or locally advanced adenocarcinoma of the exocrine pancreas (stadium UICC III/IV)
* Presence of at least one measurable (according to RECIST criteria) marker lesion (primary tumor or metastasis) outside of an area that was previously subjected to radiation therapy
* Failure of a palliative first line therapy of a metastatic or locally advanced adenocarcinoma of the exocrine pancreas due to: Progress within 3 months after a first-line therapy Discontinuation of a first-line therapy due to toxicity
* Age >= 18 years
* Karnofsky index > 60%
* Expected live span > 12 weeks
* Sufficient bone marrow reserve: Granulocytes >= 1.5 x 109/L and Platelets >= 100 x 109/L and Hemoglobin >= 9 g/L
* Serum Bilirubin < 2 x upper normal limit or 2.5 x upper normal limit in case of hepatic metastasis (biliary drainage allowed)
* AST/ALT < 2.5 x upper normal limit

Exclusion Criteria:

* Every other cancer or secondary cancer besides the basal cell carcinoma of the skin or the carcinoma in situ of the cervix uteri. Inclusion of patients with other types of cancer that were successfully treated and that did not relapse within the last 5 years is possible
* Pregnancy or lactation
* Patients able to reproduce that do not adhere to strict contraception
* Presence of brain metastasis
* Severe, uncontrolled infection
* Preexisting peripheral neuropathy > grade I
* Preexisting severe illnesses such as unstable coronary artery disease or uncontrolled cardiac arrhythmia
* Justified disbelief in the compliance of the patient
* Parallel participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
tumor response | 12/2009 and end of the study 12/2010

SECONDARY OUTCOMES:
progression free survival | 12/2009 and end of study 12/2010
overall survival | 12/2009 and end of study 12/2010
Questionnaire for quality of life | every three weeks
Questionnaire for clinical Benefit | every week
toxicity / safety | every week
  all adverse events will be documented every week with their correlation to Oxaliplatin and Docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Seufferlein, Prof. Dr., Principal Investigator — Universitätsklinikum Halle / Klinik für Innere Medizin I
Locations (5):
- Germany (5):
  - Städtische Kliniken Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Klinikum Schwäbisch Gmünd, Mutlangen, Baden-Wurttemberg
  - Universitätsklinikum Ulm Klinik für Innere Medizin I, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Giessen und Marburg GmbH, Marburg, Hesse
  - Klinik und Poliklinik für Innere Medizin I / Universitätsklinikum Halle, Halle

REFERENCES:
- [Derived] Ettrich TJ, Perkhofer L, von Wichert G, Gress TM, Michl P, Hebart HF, Buchner-Steudel P, Geissler M, Muche R, Danner B, Kachele V, Berger AW, Guthle M, Seufferlein T. DocOx (AIO-PK0106): a phase II trial of docetaxel and oxaliplatin as a second line systemic therapy in patients with advanced pancreatic ductal adenocarcinoma. BMC Cancer. 2016 Jan 15;16:21. doi: 10.1186/s12885-016-2052-4. PMID 26772812